CLINICAL TRIAL: NCT00172315
Title: Proton Magnetic Resonance Spectroscopy (1H MRS) in Evaluating the Bone Marrow, Muscle and Adipose Tissue on Normal and Human Immunodeficiency Virus Infected Subjects, With Serial Follow-Up
Brief Title: Proton Magnetic Resonance Spectroscopy (1H MRS) in Evaluating the Bone Marrow, Muscle and Adipose Tissue on Normal and Human Immunodeficiency Virus Infected Subjects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701422
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-03-29 (Estimated); Status verified 2005-08

CONDITIONS: Acquired Immunodeficiency Syndrome; Lipodystrophy
Keywords: acquired immunodeficiency syndrome; lipodystrophy; MR spectroscopy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Lipodystrophy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Magnetic resonance spectroscopy (MRS) is commonly applied in medicine with 1H proton or 31-phosphorus spectra. The proton MRS is often used in evaluating the central nervous system and 31P MRS is used in muscular diseases or neoplasms. However, the proton MRS is also considered to be applied to the musculoskeletal system because of its profound amount of protons. Ballon used the STEAM technique, and Schick used the PRESS technique, to investigate the lipid and water spectra of the bone marrow and also correlated those with hematological diseases and post-treatment effects. Schellinger et al. used the STEAM sequence to calculate the lipid content of the vertebral bone marrow and found that it was influenced according to age and sex. The investigator had used the proton MRS to evaluate the lipid and water spectra of the femoral head and revealed its significance in predicting avascular necrosis of the femoral head. According to the above research literature, the investigators considered further investigation of the proton MRS in evaluating the musculoskeletal system.

DETAILED DESCRIPTION:
Magnetic resonance spectroscopy (MRS) is commonly applied in medicine with 1H proton or 31-phosphorus spectra. The proton MRS is often used in evaluating the central nervous system and 31P MRS is used in muscular diseases or neoplasms. However, the proton MRS is also considered to be applied to the musculoskeletal system because of its profound amount of protons. Ballon used the STEAM technique, and Schick used the PRESS technique, to investigate the lipid and water spectra of the bone marrow and also correlated those with hematological diseases and post-treatment effects. Schellinger et al. used the STEAM sequence to calculate the lipid content of the vertebral bone marrow and found that it was influenced according to age and sex. The investigator had used the proton MRS to evaluate the lipid and water spectra of the femoral head and revealed its significance in predicting avascular necrosis of the femoral head. According to the above research literature, the investigators considered further investigation of the proton MRS in evaluating the musculoskeletal system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of acquired immunodeficiency syndrome (AIDS)
* Normal volunteers

Exclusion Criteria:

* AIDS patients with newly developed neoplasms

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Ting-Fang Shih, M.D., Principal Investigator — Department of Medical Imaging, National Taiwan University Hospital
Locations (1):
- Tiffany Ting-Fang Shih, Taipei, Taiwan